CLINICAL TRIAL: NCT04878757
Title: Implementing Inclusive Fraction Intervention Classwide
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Doug Fuchs, Professor Special Education, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 191312
Record Dates: First submitted 2021-04-23; First posted 2021-05-07 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Math Learning Difficulty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CFI - Classwide Fraction Intervention (Experimental): 40 sessions (2 sessions per week; 25-31 minutes per session) of explicit fraction intervention designed to improve students understanding of fraction magnitude and fraction operations.
  Interventions: Behavioral: CFI - Classwide Fraction Intervention
- Control - Business-As-Usual (No Intervention): Involves participation in the schools' typical math program

INTERVENTIONS:
Behavioral: CFI - Classwide Fraction Intervention — 40 sessions (2 sessions per week; 25-31 minutes per session) of explicit fraction intervention designed to improve students understanding of fraction magnitude and fraction operations.
  Arms: CFI - Classwide Fraction Intervention

SUMMARY:
The main purpose of this study is to assess effects of a previously validated fraction intervention when it is conducted classwide on the fraction knowledge of fourth-grade students with and without math learning difficulties (MLD). The study population is 4th-grade students with MLD and without MLD. Teachers agree to be randomly assigned to two conditions. In one condition, teachers include classwide fraction intervention (CFI) in their standard math program. In the other condition, teachers conduct their standard math program without CFI. CFI is implemented 2 times per week for 20 weeks for about 30 minutes each time. Students in both conditions are tested before and after CFI ends.

DETAILED DESCRIPTION:
The study is conducted in the Metropolitan-Nashville Public Schools. Teachers decide if they want to participate. Parents of students in their classrooms decide if they want their children to participate in the study; participation means students complete the study's pretesting and posttesting, and teachers report their test scores on a school-collected measure. Students decide if they want to participate. Teachers complete a survey, report student scores on the school-collected measure, and are observed during CFI implementation.

Each CFI session comprises 3 segments. In Segment 1 (10-12 minutes), teachers conduct that day's CFI lesson. In Segment 2 (10-12 minutes), students work in pairs, taking turns being "coach" and "player" as they explain their thinking and solution strategies taught in that day's Segment 1. Students use CFI help cards to provide constructive feedback to each other. Segment 3 (5-7 minutes) is independent practice.

The primary end-points are students' posttest fraction ordering, fraction number line estimate, fraction calculations. Secondary end-points are students' performance on more distal fraction measures. Other measures are a teacher survey describing fractions instruction and reliance on CFI procedures and their perceptions of CFI's effectiveness and feasibility, as well as CFI adherence from audio recordings and live observations of teachers implementing CFI.

ELIGIBILITY:
Inclusion Criteria:

* To enter the study, students must meet the following criteria. They must attend a Metropolitan-Nashville Public School whose principal has given permission for his/her school to participate and participate in a fourth-grade classroom whose teacher has agreed to let her/his students participate.

Exclusion Criteria:

* We exclude students with identified intellectual disability from study data collection because CFI is not designed to meet the needs of this population. There are no other exclusions.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2210 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fraction Ordering Score | Pre-intervention measurement will take place within three weeks prior to beginning of intervention; post-intervention measurement will take place within three weeks after completion of intervention.
  In Fraction Ordering, students order 11 strings of 3 fractions to be ordered from least to greatest. The student's score is the change from pre-intervention to post-intervention in the number of correctly ordered strings.
Change in Fraction Number Line Estimation Score | Pre-intervention measurement will take place within three weeks prior to beginning of intervention; post-intervention measurement will take place within three weeks after completion of intervention.
  In Fraction Number Line Estimation, students place fractions on a 0-2 number line, presented via computer with labeled endpoints. Accuracy for each of the 20 items is the absolute value of the difference between actual and correct answer multiplied by 100. The student's score is the change from pre-intervention to post-intervention in average accuracy across all 20 items.
Change in Fraction Calculations Score | Pre-intervention measurement will take place within three weeks prior to beginning of intervention; post-intervention measurement will take place within three weeks after completion of intervention.
  In Fractions Calculations, students complete 25 fraction calculation problems with like and unlike denominators, with and without whole or mixed numbers. The student's score is the change from pre-intervention to post-intervention in the number of correct answers.

SECONDARY OUTCOMES:
Change in Fraction Arithmetic Number Line Estimation Score | Pre-intervention measurement will take place within three weeks prior to beginning of intervention; post-intervention measurement will take place within three weeks after completion of intervention.
  In Fraction Arithmetic Number Line Estimation, students estimate placement of the total or difference of 16 fraction addition and subtraction problems on number lines. Accuracy for each of the items is the absolute value of the difference between actual and correct answer multiplied by 100. The student's score is the change from pre-intervention to post-intervention in the average accuracy across all items.
National Assessment of Educational Progress (NAEP) Released Fraction Items - Updated | Measurement will take place within three weeks after the end of intervention
  Students complete 12 items from the 4th-grade assessment and 8th-grade assessment, tapping fractions magnitude understanding, part-whole understanding, and fractions calculations. The student's score is the number of correct answers.
Change in Fraction Magnitude & Calculations in Context Score | Pre-intervention measurement will take place within three weeks prior to beginning of intervention; post-intervention measurement will take place within three weeks after completion of intervention.
  In Fraction Magnitude and Calculations in Context, students complete 14 word problems: 3 involving ordering, 3 involving making units into fractions, and 8 involving additional and subtraction to reflect a change in quantity over time. The student's score is the change from pre-intervention to post-intervention in the number of problems answered correctly.
Measures of Academic Progress (MAP) | Within six weeks of intervention completion
  These scores are students' scores on the school district's Northwest Evaluation Association Measures of Academic Progress (NWEA MAP) testing for Numbers and Operations as reported by classroom teachers. Percentile scores range from 0 to 99. The Rasch Unit (RIT) scores range from 100-300. For both measures, higher scores indicate a better outcome.

OTHER OUTCOMES:
Fall Teacher Survey | 4-6 weeks after intervention begins
  In a structured survey, teachers describe their methods for teaching fractions and their reliance on CFI's design dimensions. Teachers rate the accuracy of statements using a 1-5 scale and distribute 100 points to indicate their instructional emphasis. Descriptive statistics for each item on the survey are reported (rating score or percentage of points allocated).
Spring Teacher Survey | 14-16 weeks after intervention begins
  In a structured survey, teachers describe their methods for teaching fractions and their reliance on CFI's design dimensions. Teachers rate the accuracy of statements using a 1-5 scale and distribute 100 points to indicate their instructional emphasis. Descriptive statistics for each item on the survey are reported (rating score or percentage of points allocated).

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Fuchs, Ph.D., Principal Investigator — Vanderbilt University
Locations (1):
- Metropolitan Nashville Public Schools, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make de-identified datasets electronically available to external users under a signed data-sharing agreement (see Access Criteria). The outside user submits a request describing the variables of interest and the research design. If approved, a Data Use Agreement Form will be sent to the user to complete. If approved, the relevant dataset data will be extracted and provided with relevant portions of the data dictionary. If not, written communication will be provided explaining the basis for this decision. If we are unclear, a written request for clarifications will be provided, with up to two rounds of clarifications.
Time Frame: Variables will become available as manuscripts reporting those variables are accepted for publication. The PI will respond within 2 months to an external user's request that describes the external user's variables of interest and research plan,
Access Criteria: The proposed variables are part of the database; the research questions can be answered with those variables; & the research plan is internally consistent, quantitatively sound, and tenable. Also, guarantees are provided that data are used only for the research purposes described in the user's request; no individual will be identified for any purpose; the data will be secured appropriately; the data will be destroyed or returned after analyses are completed; a written research report will be provided to the PI (or her designee) within 12 months of receiving the database; and the user will cite the parent study in all presentations, written reports, & publications.

DOCUMENTS (1):
  • Informed Consent Form (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT04878757/ICF_000.pdf